CLINICAL TRIAL: NCT01394445
Title: Influence of Physostigmine on Patient-Controlled Analgesia
Brief Title: Pilot Study of Physostigmine-Enhanced Opioid Analgesia
Acronym: PHANOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-510ex09/10; 2010-021901-19 (EudraCT Number)
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Physostigmine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physostigmine (Active Comparator)
  Interventions: Drug: Physostigmine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Physostigmine — continuous intravenous infusion per syringe pump (13 vials of 2 mg/5 ml --> 26 mg/65 ml; 1 ml = 0.4 mg Physostigmine) at rate of 1 mg/h (2.5ml/h) for 24 hours
  Arms: Physostigmine
Drug: Placebo — continuous intravenous infusion of 65 ml NaCl 0.9% with syringe pump at rate of 2.5 ml/h for 24 hours
  PCA: Patient-controlled analgesia with hydromorphone 0.2 mg/ml, on demand: bolus of 0.2 mg, maximum 5 boli per hour; 4-hour-maximum 4 mg
  Other Names: sodium chloride; hydal
  Arms: Placebo

SUMMARY:
The investigators hypothesize that the administration of physostigmine in the postoperative period after nephrectomy reduces opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* At least 50 kg
* Suitable for PCA
* ASA 1-3

Exclusion Criteria:

* Bronchial asthma/severe or exacerbated COPD
* Iritis
* Stenoses/spasms of intestine, urinary tract, biliary tract
* Closed traumatic brain injury
* Severely reduced left ventricular function (EF<30%)
* Recent myocardial infarction
* Recent stroke
* Known allergy or hypersensitivity or contraindications against hydromorphone, physostigmine
* History of alcohol or drug abuse
* Patients enrolled in another study
* Women of childbearing age without a negative pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
opioid consumption | 24 hours

SECONDARY OUTCOMES:
pain scores | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Rumpold-Seitlinger, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Hospital of the Medical University of Graz, Graz, Styria, Austria